CLINICAL TRIAL: NCT06084104
Title: A Phase 1, Single-Dose, Non-Randomized, Open Label Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of DZD9008
Brief Title: DZD9008 PK Study in Hepatic Impairment Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Collaborators: PPD Development, L.P. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZ2022E0007
Record Dates: First submitted 2023-09-06; First posted 2023-10-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hepatic impairment (Experimental): Subjects with hepatic impairment
  Interventions: Drug: DZD9008
- Healthy Subject (Experimental): Subjects with normal hepatic function
  Interventions: Drug: DZD9008

INTERVENTIONS:
Drug: DZD9008 — A single oral dose of 200mg DZD9008
  Arms: Hepatic impairment
Drug: DZD9008 — A single oral dose of 200mg DZD9008
  Arms: Healthy Subject

SUMMARY:
This study will investigate the pharmacokinetics, safety, and tolerability of DZD9008 in subjects with hepatic impairment compared to subjects with normal hepatic function

ELIGIBILITY:
Inclusion criteria:

1. The subject is male or female 18 to 75 years of age, inclusive, at screening.
2. The subject has a BMI of 18.0 to 40.0 kg/m2, inclusive, at screening and check-in.
3. The subject has a minimum body weight of 50.0 kg, at screening and check-in.
4. The subject has a resting pulse rate of ≥ 40 and < 100 beats per minute with no clinically significant deviation as judged by the investigator.
5. The subject agrees to comply with all protocol requirements.
6. The subject is able to provide written informed consent.

   Additional Inclusion Criteria for Healthy Subjects Only (Cohort 2) Only (7-11):
7. The subject has normal hepatic function. No known or suspected hepatic impairment based on liver function tests (e.g., ALT, AST, ALP, and bilirubin), albumin, and prothrombin time is defined as the following with a single repeat permitted to assess eligibility if needed, at screening and check-in:

   1. ALT and AST ≤ ULN
   2. Total bilirubin ≤ ULN (subjects with a history of Gilbert syndrome are eligible if they only have elevated total bilirubin)
   3. ALP ≤ ULN
   4. Albumin ≥ 3.6 g/dL
   5. Prothrombin time ≤ ULN
8. The subject has a resting blood pressure of 90 to 145 mmHg (systolic) and 40 to 95 mmHg (diastolic), at screening and check-in.
9. The subject has a QTcF of ≤ 450 msec, at screening and check-in.
10. The subject is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12 lead ECG results, and physical examination findings.
11. Each subject with normal hepatic function (Cohort 2) must individually match a subject with impaired hepatic function (Cohort 1) by age (± 10 years), body weight (± 10 kg), and sex (similar distribution of males and females).

    Additional Inclusion Criteria for Subjects with Hepatic Impairment (Cohort 1) Only (12-18):
12. The subject satisfies the Class B of the Child-Pugh classification (no albumin use within 14 days). Six out of 10 subjects also meet NCI ODWG Group C criteria.
13. The subject has a diagnosis of hepatic dysfunction due to hepatocellular disease (and not secondary to any acute ongoing hepatocellular process), with features of cirrhosis due to any etiology, except for DILI, which is confirmed by at least one of the following criteria:

    1. histologically by prior liver biopsy showing cirrhosis
    2. clinically by physical examination, laboratory data, liver imaging, or endoscopic findings
14. The subject has following clinical laboratory values, at screening and check-in:

    1. ALT and AST ≤ 5 × ULN
    2. Total bilirubin ≤ 3 × ULN
    3. ANC ≥ 1.5 × 109/L
    4. Platelet count ≥ 30 × 109/L
    5. Hemoglobin ≥ 90 g/L
15. The subject has chronic (more than 6 months) and stable hepatic impairment (ie, no acute episodes of illness within 30 days before screening due to deterioration of hepatic function) as assessed by the NCI-ODWG criteria (Group C) or a Child-Pugh classification score of moderate (7 to 9 points).
16. The subject has a resting blood pressure of 90 to 155 mmHg (systolic) and 50 to 100 mmHg (diastolic), at screening and check-in.
17. The subject has a QTcF of ≤ 470 msec, at screening and check-in.
18. The subject is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12 lead ECG results, and physical examination findings, except for findings that, as judged by the investigator, are consistent with the subject's hepatic impairment or other stable concomitant medical conditions.

Exclusion criteria:

1. The subject has a history or clinical manifestations of a significant neurological, renal, cardiovascular, gastrointestinal, pulmonary, hematologic, immunologic, or psychiatric disease that would preclude study participation, as judged by the investigator.
2. The subject has any surgical or medical condition that may alter the absorption, distribution, metabolism, or excretion of drugs (e.g., gastrectomy).
3. The subject has a history of cancer (malignancy) with the following exceptions:

   1. adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix, or
   2. other malignancies which have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study
4. The subject has a history of being immunocompromised or has a positive test result for HIV types 1 or 2 antibodies at screening.
5. The subject has an acute or chronic infection requiring treatment with oral antibiotics (except, rifaximin for the treatment of hepatic encephalopathy), antivirals, antiparasitic, antiprotozoals, or antifungals within 4 weeks prior to Day 1 or superficial skin infection within 1 week prior to Day 1.
6. The subject has a history of risk factors for Torsades de Pointes (e.g., heart failure/cardiomyopathy or family history of long QT syndrome), has clinically significant hypokalemia or hypomagnesemia, and is taking concomitant medications that prolong the QT/QTc interval.
7. The subject has uncontrolled hypertension despite optimal medical management.
8. The subject had arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study drug administration.
9. The subject tests positive for breath alcohol test at screening and on check-in (Day 1).
10. The subject is unable or unwilling to restrict smoking to 5 cigarettes or less per day.
11. The subject is involved in strenuous activity or contact sports within 24 hours of the first dose of study drug or during the study.
12. The subject has donated blood (excluding plasma donation) of ≥ 500 mL within 60 days before the first dose of study drug.
13. The subject has poor peripheral venous access.
14. The subject should not be any of the following:

    1. investigator staff member or their family members
    2. site staff member otherwise supervised by the investigator, or employees, including their family members, directly involved in the conduct of the study
15. The subject has a history of relevant drug and/or food allergies (ie, allergy to DZD9008 or any excipients, or any significant food allergy).
16. The subject has received DZD9008 or any other investigational drug in another investigational study within 30 days of dosing.
17. The subject is enrolled in another clinical study or has used any investigational drug or device within 4 weeks (or 5 times the half-life of the pervious drug [if known], whichever is longer), prior to dosing with study drug. The window will be derived from the date of the last dose of study drug in the previous study.
18. The subject has used a strong or moderate inhibitor or inducer of CYP3A4 and/or P gp including St. John's Wort, within 14 days and 28 days, respectively, prior to dosing and until the completion of the last PK sample collection unless it is deemed acceptable following consultation with Dizal Pharma's medical monitor and the investigator.
19. The subject has used PPIs within 5 days prior to dosing until 24 hours after dosing. Use of H2-antagonists and antacids within 12 hours prior to dosing until 12 hours after dosing unless it is deemed acceptable following consultation with Dizal Pharma's medical monitor and the investigator.
20. In the opinion of the investigator, the subject is not suitable for entry into the study.

    Additional Exclusion Criteria for Healthy Subjects Only (Cohort 2):
21. The subject with normal hepatic function has any of the following:

    1. evidence or history of bleeding diathesis, or
    2. any hemorrhage or moderate bleeding event within 4 weeks of start of study drug administration
22. The subject has a positive result for HBsAg or HCV Ab.
23. The subject has an estimated glomerular filtration rate (CKD-EPI formula or Cockcroft-Gault method) of < 90 mL/min.
24. The subject has used any vaccine or used any prescription (excluding hormonal birth control and hormone replacement therapy) or over the counter medications (except paracetamol [up to 2 g per day]), including herbal or nutritional supplements, within 14 days before the first dose of study drug and throughout the study.
25. The subject has a positive test result for drugs of abuse or alcohol at screening or before the first dose of study drug.

    Additional Exclusion Criteria for Subjects with Hepatic Impairment Only (Cohort 1):
26. The subject has fluctuating or rapidly deteriorating hepatic function, as indicated by recent history or worsening of clinical (ie, abdominal pain, nausea, vomiting, anorexia, or fever) and/or laboratory signs of hepatic impairment, as judged by the investigator.
27. The subject has evidence of acute viral hepatitis within 30 days before dosing with study drug.
28. The subject has an active hepatitis B or C viral infection.
29. The subject has history or symptoms of hepatic encephalopathy Grade 2 or above within 3 months prior to screening visit.
30. The subject has a history of unstable diabetes mellitus as evidenced by HbA1c ≥ 9% at screening.
31. In the opinion of the investigator, the subject has clinically demonstrable severe ascites and/or pleural effusion.
32. The subject has evidence of hepatopulmonary syndrome, hydrothorax, or hepatorenal syndrome.
33. The subject had an organ transplant or is on a waiting list.
34. The subject had a portosystemic shunt (including transjugular intrahepatic portosystemic shunts).
35. The subject has an estimated glomerular filtration rate (CKD-EPI formula) of < 60 mL/min.
36. The subject has symptoms consistent with spontaneous bacterial peritonitis, known active spontaneous bacterial peritonitis, or a history of spontaneous peritonitis within the last 6 months.
37. The subject is suspected of having hepatocellular carcinoma (ie, if α fetoprotein > 50 ng/mL at screening), subjects will undergo appropriate diagnostic studies (e.g., CT scan or hepatic ultrasound) to exclude the possibility of hepatocellular carcinoma.
38. The subject has received any vaccine or used any prescription (excluding hormonal birth control and hormone replacement therapy) or over the counter medications, including herbal or nutritional supplements, within 14 days before the first dose of study drug and throughout the study, except those essential for the management of hepatic impairment or the treatment of stable concomitant medical conditions, as judged by the investigator. The dose of an approved medication must remain stable from 7 days before study drug dosing and throughout the study.
39. The subject has a positive test result for drugs of abuse (except positive test results associated with prescription medications that have been reviewed and approved by the investigator) or alcohol at screening or prior to study drug dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma (peak) drug concentration [Cmax] | Day 1 to day 14
Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 to day 14
Area under the plasma concentration-curve from time zero to last quantifiable concentration (AUClast) | Day 1 to day 14

SECONDARY OUTCOMES:
Apparent total body clearance (CL/F) | Day 1 to day 14
Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 to day 14
Terminal phase half-life (t1/2), | Day 1 to day 14
Time to maximum observed plasma concentration (Tmax) | Day 1 to day 14
Fraction unbound (Fu) | Day 1 to day 14
Unbound area under plasma concentration time curve from zero to infinity (AUC0-inf, u) | Day 1 to day 14
Unbound area under the plasma concentration-curve from time zero to last quantifiable concentration (AUC0-last, u) | Day 1 to day 14
Unbound maximum observed plasma (peak) drug concentration (Cmax, u) | Day 1 to day 14
Unbound apparent total body clearance (CLu/F) | Day 1 to day 14
Unbound apparent volume of distribution (Vz,u/F) | Day 1 to day 14
Adverse events | Day 1 to day 14
Clinical laboratory test results: hematology, coagulation, serum chemistry, urinalysis | Day 1 to day 14
12-lead ECG results: tracings, rhythm, RR interval, PR interval, QRS width, QT interval, and QTcF | Day 1 to day 14
Vital sign measurements: systolic and diastolic blood pressure, pulse rate, respiratory rate and body temperature | Day 1 to day 14
Physical examination findings: assessment of skin, head, ears, eyes, nose, throat, neck, thyroid, lungs, heart, cardiovascular, abdomen, lymph nodes, and musculoskeletal system/extremities | Day 1 to day 14

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Marbury, MD, Principal Investigator — Orlando Clinical Research Center; Eric Lawitz, MD, Principal Investigator — Texas Liver Institute
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation, San Antonio, Texas